CLINICAL TRIAL: NCT03174834
Title: Bladder Stimulation Technique for Clean Catch Urine Collection in Infants : Assessing Impact on Patients and Providers in a Pediatric Emergency Department
Brief Title: Bladder Stimulation Technique for Clean Catch Urine Collection in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Michigan (Other)
Collaborators: Sarnaik Endowment Fund (Unknown); CHMF Annual Fund (Unknown); Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Yagnaram Ravichandran, MBBS, MD, FAAP, Fellow, Pediatrics Emergency Medicine, Children's Hospital of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1702000315
Record Dates: First submitted 2017-05-27; First posted 2017-06-05 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Urinary Tract Infections
Keywords: Bladder Stimulation Technique; Clean Catch Urine; UTI in infants less than 6 months
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bladder Stimulation Technique (Other): Single arm study, where urine collection will be done via bladder stimulation and subsequently catheterization if they meet the eligibility criteria.
  Interventions: Other: Bladder Stimulation technique

INTERVENTIONS:
Other: Bladder Stimulation technique — The bladder stimulation technique is performed following genital cleaning with a 2% castile soap towelette, which is part of the sterile clean catch urine collection cup kit. For the technique, infants will be held under their armpits by a parent over the bed, with legs dangling in males and hips flexed in females. The nurse or technician will then alternate between bladder stimulation maneuvers: gentle tapping in the suprapubic area at a frequency of 100 taps per minute for 30 seconds followed by lumbar paravertebral massage maneuvers for 30 seconds. These two stimulation maneuvers will be repeated until micturition begins, or for a maximum of 300 seconds.

SUMMARY:
Urinary tract infection is the most common serious bacterial infection among infants. Bladder catheterization is considered the gold standard for diagnosis, yet is painful and invasive. In contrast, the bladder stimulation technique has been shown to be a quick and non-invasive approach to collecting urine in young infants with a contamination rate similar to bladder catheterization. Previous research, however, relied upon trained study personnel thereby limiting the generalizability of their findings. By training staff in the pediatric emergency department, this study aims to evaluate the feasibility of incorporating this technique into routine clinical practice while also assessing its impact on parent and provider satisfaction.

DETAILED DESCRIPTION:
Previous studies have demonstrated that the bladder stimulation technique is a quick and non-invasive approach to collecting urine in young infants with a contamination rate similar to the current more invasive gold standard, catheterization. This study, however, will be the first to demonstrate the feasibility of incorporating this technique into clinical practice in a busy, urban, academic pediatric emergency department (PED). In training over 120 PED staff, the investigators aim to demonstrate that minimal training is required to perform this technique. In addition, the investigators hypothesize that the bladder stimulation technique will be well tolerated by patients, and preferred by providers and parents when compared with catheterization. The results of this study may then lead to a change in practice where the bladder stimulation technique will be used preferentially for infants requiring a urinalysis and urine culture.

Urinary tract infection (UTI) is the most common serious bacterial infection among febrile infants, occurring in 7% of children less than 24 months of age evaluated for fever without a source. The American Academy of Pediatrics (AAP) recommends obtaining a urine specimen for urinalysis and culture via suprapubic aspiration (SPA) or catheterization, particularly for infants requiring immediate antimicrobial therapy. These methods are painful and invasive, yet are considered the gold standard approaches to urine collection in infants as the culture obtained has a sensitivity and specificity of >95%. Alternative techniques, such as a urine collection bag attached to the perineum or a clean catch urine (CCU), offer non-invasive approaches to urine collection but are undesirable as cultures obtained using a bag have a false positive rate approaching 90% and CCU can be time consuming. As an alternative to these methods, Herreros et al described a new non-invasive technique for obtaining a mid-stream CCU sample in newborns. This approach couples feeding with bladder stimulation and was successful in 86% of newborns with a mean time of 57 seconds. Subsequent research has demonstrated that this technique is particularly effective for children ≤ 90 days with a contamination rate similar to that of catheterization. While previous studies have demonstrated the ease of this approach, without an increase in contamination rates compared with more invasive techniques, previous studies have relied upon trained study personnel, limiting the generalizability of the technique.

The proposed study builds upon published literature. Herreros et al first described the bladder stimulation technique in newborn infants, which was successful in 86% of newborns with a mean time of 57 seconds. Altuntas et al subsequently demonstrated in a randomized controlled study that the bladder stimulation technique was effective in 78% of newborns, with urine collection occurring within a median time of 60 seconds. Tran et al then demonstrated that this technique is particularly effective for children ≤ 90 days presenting to the emergency department with a contamination rate similar to that of catheterization. Importantly, these findings were replicated by Labrosse et al who also noted that the contamination proportion is not statistically different from the rate seen with catheterization. Thus, while all the previous studies have demonstrated the ease of this approach, without an increase in contamination rates compared with more invasive techniques, previous studies have relied upon trained study personnel, limiting the generalizability of the technique to routine clinical care.

This study will be conducted in the PED at the Children's Hospital of Michigan, an academic tertiary care facility in an inner city setting with approximately 90,000 PED visits annually.

The investigators estimate a sample size of 92 patients to be recruited over the study period. This was based on a margin of error (e=0.10) obtained from the study by Labrosse et al. The investigators estimate a success rate of 40% for the bladder stimulation technique, with a 5% level of significance (p < 0.05).

Following informed consent, demographic data will be obtained by a trained research assistant using a standardized form. The bladder stimulation technique will be performed by a trained PED nurse or technician using the procedure outlined below. Prior to the six month period of patient recruitment, all technicians and nursing staff in the PED will receive standardized training using a video module and print materials. The steps of the procedure will also be printed and available in the PED as reference material. The bladder stimulation technique will adhere to the protocol previously published by Herreros et al and replicated by Labrosse et al. The technique involves a combination of fluid intake and noninvasive bladder stimulation maneuvers. All infants will be encouraged to feed during a 20-minute period prior to the stimulation technique. Breast fed infants will feed ad libitum whereas formula fed infants will be offered an age and weight appropriate volume (1 day of age 10 ml; 2 - 7 days of age, add 10 ml / day of life to a maximum of 70 ml / feed; ≥ 8 days of age 25 mg / kg of formula). Infants who do not feed well will not be excluded. Infants who are determined to need intravenous fluids at the discretion of the treating physician will receive a standard 10-20 ml / kg bolus of normal saline over < 30 minutes. Specimen collection using the bladder stimulation technique will be started 20 minutes after the initiation of oral feeding and/or intravenous fluids.

The bladder stimulation technique is performed following genital cleaning with a 2% castile soap towelette, which is part of the sterile clean catch urine collection cup kit. For the technique, infants will be held under their armpits by a parent over the bed, with legs dangling in males and hips flexed in females. The nurse or technician will then alternate between bladder stimulation maneuvers: gentle tapping in the suprapubic area at a frequency of 100 taps per minute for 30 seconds followed by lumbar paravertebral massage maneuvers for 30 seconds. These two stimulation maneuvers will be repeated until micturition begins, or for a maximum of 300 seconds. The nurse or technician performing the bladder stimulation technique or a resident or medical student caring for the patient will collect the urine in a clean catch specimen container. The research assistant will time the procedure from the start of the stimulation techniques to the start of micturition using a stopwatch. In accordance with current PED practices for pain control, non nutritive sucking on a pacifier with/without sucrose will be provided as an optional comfort measure, based on parental preference.

Urine will be sent to the laboratory for urinalysis and culture in accordance with standard laboratory techniques. Failure to obtain a specimen after continued bladder stimulation maneuvers for > 300 seconds will necessitate obtaining a catheterized urine sample. When catheterization is required, this will be obtained by a technician or nursing staff in accordance with their established protocols for this procedure. To preserve the current standard of care, catheterization or SPA will also be performed when: (1) the urinalysis obtained using the bladder stimulation technique is positive and/or (2) the treating physician decides to prescribe antibiotics. Catheterization may also be performed at the discretion of the treating physician. When catheterization is performed, the research assistant will time the procedure from the start of catheter placement to urine collection using a stopwatch. In accordance with current PED practices for pain control, non nutritive sucking on a pacifier with/without sucrose will also be provided for this procedure as an optional comfort measure, based on parental preference.

During the bladder stimulation technique, parental perception of pain will be assessed using the Numeric Rating Scale (NRS). The research assistant will administer the NRS to the parent immediately prior to the procedure (T0), during the bladder stimulation technique (T1), 1 minute after completion of the bladder stimulation technique (T2) and 5 minutes after completion of the bladder stimulation technique (T3). For infants undergoing catheterization, parental perception of pain will also be assessed using the NRS at similar time intervals.

After collection of the urine sample using the stimulation technique (whether successful or not), the parent and the nurse will complete a brief questionnaire (administered by the research assistant). The parent questionnaire aims to evaluate parental perception of discomfort and their satisfaction with the stimulation technique. The provider questionnaire evaluates their comfort with the procedure and their perception of patient discomfort. Similar questionnaires will be distributed to the parent and the nurse following catheterization when this procedure is performed. Following the clinical encounter, the research assistant will review participants' electronic medical record to obtain the final results of the urinalysis and urine culture to complete the standardized data collection form for the participant.

A successful urine specimen obtained using the bladder stimulation technique will be defined by the collection of at least 1 mL of urine within 300 seconds of initiating the bladder stimulation maneuvers. Laboratory definitions of a positive urinalysis and urine culture are defined below based on definitions published by the American Academy of Pediatrics and previous authors investigating the bladder stimulation technique. As per Labrosse et al, poor oral intake will be defined as <25% of regular fluid intake during the feeding period prior to the bladder stimulation technique, based on parental assessment. Finally, the cost of the procedures (invasive versus non-invasive) will be based on the cost of material required for a clean catch urine specimen versus the cost of material required for bladder catheterization.

ELIGIBILITY:
Inclusion Criteria:

- Infants less than 6 months of age who require a urine sample for urinalysis and culture as part of their PED visit (as determined by the treating physician) are eligible for inclusion

Exclusion Criteria:

* Parents / caregivers do not speak English
* Parents / guardian unavailable to sign consent
* Evidence of injury / infection to the abdomen / back precluding completion of the bladder stimulation technique
* Known medical condition rendering it impossible to obtain a sample using the stimulation technique (e.g. urostomy)
* Critical illness and/or hemodynamic instability
* Current antibiotic therapy or antibiotics within 14 days of enrollment
* Previous enrollment.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom urine collection is successful using the bladder stimulation technique | 6 Months
  The technique will be performed following genital cleaning. Infants will be held under their armpits by a parent over the bed, with legs dangling in males and hips flexed in females followed by gentle tapping in the suprapubic area at a frequency of 100 taps per minute for 30 seconds followed by lumbar paravertebral massage maneuvers for 30 seconds. These two stimulation maneuvers will be repeated until micturition begins, or for a maximum of 300 seconds. Urine will be collected in a clean catch specimen container. The research assistant will time the procedure from the start of the stimulation techniques to the start of micturition using a stopwatch. Non nutritive sucking on a pacifier with/without sucrose will be provided as an optional comfort measure. A successful urine collection using the bladder stimulation techniques will be defined by onset of micturition within 300 seconds of bladder stimulation.
Proportion of bacterial contamination among samples collected using the bladder stimulation technique | 6 months
  Contamination rates of urine cultures obtained using the bladder stimulation technique will be expressed in terms of proportion to the total sample size and this rate will be compared to the contamination rates of urine cultures obtained via catheterization.
  The criteria for contamination will be determined per the AAP guidelines for positive urine culture versus contamination rates.
  Laboratory definitions of a positive urinalysis and urine culture are defined based on definitions published by the American Academy of Pediatrics and previous authors investigating the bladder stimulation technique.
  * Three criteria are needed for each definition: Urinalysis result, number of organisms cultured and specific threshold for colony counts based on method of collection.
  * Positive urinalysis: Bacteriuria, positive leukocyte esterase test, positive nitrite test and/or >/= 10 white blood cells per micro liter; negative urinalysis: do not meet criteria for positive urinalysis

SECONDARY OUTCOMES:
Time required for successful urine collection using the bladder stimulation technique | 6 Months
  The investigators aim to evaluate the time required for successful urine collection using the bladder stimulation technique.
  The research assistant will time the procedure from the start of the stimulation techniques to the start of micturition using a stopwatch. The timing will start from the time the bladder stimulation maneuvers start after the patient is positioned and cleaned till the onset of micturition or until 300 seconds, whichever is earlier. The investigators aim to assess the time taken for successful urine collection using bladder stimulation, especially since prior studies have reported onset of urination within 57 seconds. the ultimate goal is to show that this method of collection is easy, minimally invasive and quick.
Time required for successful urine collection from the start of feeding | 6 Months
  The investigators also aim to evaluate the time required for successful urine collection for the entire bladder stimulation technique (initiation of feeding to start of voiding). The research associate will retrospectively review charts and look at the time feeding was initiated and the time taken till the onset of micturition. By doing this, the investigators aim to evaluate the total time of the procedure and thereby establish this as a potentially rapid and quick procedure as compared to catheterization with potential impact on the length of stay.
Patient distress ( parental perception ) during bladder stimulation technique | 6 Months
  The investigators aim to evaluate patient distress during the bladder stimulation technique using the Numeric Rating Scale (NRS).
  During the bladder stimulation technique, parental perception of pain will be assessed using the Numeric Rating Scale (NRS). The research assistant will administer the NRS to the parent immediately prior to the procedure (T0), during the bladder stimulation technique (T1), 1 minute after completion of the bladder stimulation technique (T2) and 5 minutes after completion of the bladder stimulation technique (T3). For infants undergoing catheterization, parental perception of pain will also be assessed using the NRS at similar time intervals.
Parent and provider satisfaction with bladder stimulation technique | 6 Months
  The investigators aim to evaluate parent and provider satisfaction with urine collection using the bladder stimulation technique.
  After collection of the urine sample using the stimulation technique (whether successful or not), the parent and the nurse will complete a brief questionnaire (administered by the research assistant). The parent questionnaire aims to evaluate parental perception of discomfort and their satisfaction with the stimulation technique. The provider questionnaire evaluates their comfort with the procedure and their perception of patient discomfort. Similar questionnaires will be distributed to the parent and the nurse following catheterization when this procedure is performed.
Economic impact of the bladder stimulation technique | 6 Months
  The investigators aim to evaluate the economic impact of the bladder stimulation technique.
  The cost of the bladder stimulation technique will be based on cost of the urine collection cup and nursing time spent on the maneuver. This will be compared to the cost of a urine catheterization kit. Ultimate aim is to evaluate and establish bladder stimulation clean catch as a more cost effect method compared to catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Yagnaram Ravichandran, MD, Principal Investigator — Childrens Hospital of Michigan
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subcommittee on Urinary Tract Infection, Steering Committee on Quality Improvement and Management; Roberts KB. Urinary tract infection: clinical practice guideline for the diagnosis and management of the initial UTI in febrile infants and children 2 to 24 months. Pediatrics. 2011 Sep;128(3):595-610. doi: 10.1542/peds.2011-1330. Epub 2011 Aug 28. PMID 21873693
- [Background] Shaikh N, Morone NE, Bost JE, Farrell MH. Prevalence of urinary tract infection in childhood: a meta-analysis. Pediatr Infect Dis J. 2008 Apr;27(4):302-8. doi: 10.1097/INF.0b013e31815e4122. PMID 18316994
- [Background] Davies P, Greenwood R, Benger J. Randomised trial of a vibrating bladder stimulator--the time to pee study. Arch Dis Child. 2008 May;93(5):423-4. doi: 10.1136/adc.2007.116160. Epub 2008 Jan 11. PMID 18192318
- [Background] Weisz DJ, McInerney J. An associative process maintains reflex facilitation of the unconditioned nictitating membrane response during the early stages of training. Behav Neurosci. 1990 Feb;104(1):21-7. doi: 10.1037//0735-7044.104.1.21. PMID 2317278
- [Derived] Ravichandran Y, Parker S, Farooqi A, DeLaroche A. Bladder Stimulation for Clean Catch Urine Collection: Improved Parent and Provider Satisfaction. Pediatr Emerg Care. 2022 Jan 1;38(1):e29-e33. doi: 10.1097/PEC.0000000000002524. PMID 34475366